CLINICAL TRIAL: NCT00436176
Title: The Expanded Chronic Care Model: Targeting Disparities in Diabetes Care
Brief Title: Improving Diabetes Care for African Americans
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard Vanguard Medical Associates (Other)
Collaborators: Brigham and Women's Hospital (Other); Harvard University (Other)
Responsible Party: Thomas Sequist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 59751
Record Dates: First submitted 2007-02-14; First posted 2007-02-16 (Estimated); Last update posted 2009-03-23 (Estimated); Status verified 2009-03

CONDITIONS: Diabetes
Keywords: Diabetes mellitus; Quality of Health Care; Cultural Competency; Performance Feedback; Health navigator; Health disparities; Racial disparities
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intervention clinicians receive monthly performance reports, cultural competency training, and health navigation training
  Interventions: Behavioral: Expanded Chronic Care Model
- 2 (No Intervention): Control clinicians function within the context of the generic chronic care model.

INTERVENTIONS:
Behavioral: Expanded Chronic Care Model — Intervention clinicians receive monthly performance feedback reports, cultural competency training, and health navigation training.
  Arms: 1

SUMMARY:
The goal of this study is to investigate methods of improving diabetes care for African Americans in primary care clinics. Primary care clinicians will receive training in the delivery of cross-cultural medicine as well as regular performance feedback reports.

DETAILED DESCRIPTION:
Effective solutions are needed to address the parallel persistence of a quality chasm and racial disparities in diabetes care. Many large health care systems are adopting components of the Chronic Care Model to achieve substantial gains in diabetes care, though few health systems have successfully incorporated elements specific to minority health. We have previously identified racial disparities in key diabetes outcomes measures within an integrated health care delivery system, Harvard Vanguard Medical Associates (HVMA). This project will use a randomized, controlled study design within HVMA to evaluate whether enhancements to the Chronic Care Model can produce significant improvement in the quality of diabetes care for black patients. Intervention clinicians will receive monthly panel-level disparities report cards, health navigation training, and cultural competency training, while control clinicians will function within the context of the generic Chronic Care Model. The study will occur over a 12 month period and involve 4,000 white patients and 2,500 black patients with diabetes receiving care at 8 health centers. The primary outcomes will include rates of glucose (HbA1c <7.0), LDL cholesterol (<100 mg/dL), and blood pressure (<130/80) control. We will use patient focus groups to identify significant barriers to care and guide health navigation training. We will survey clinicians pre- and post intervention to assess the effect of the intervention on knowledge and attitudes towards disparities. Patient experiences will be assessed pre- and post-intervention using a validated instrument to determine whether the intervention can reduce existing racial disparities in patient reports of quality. We will perform a cost analysis related to the intervention using a health system perspective. In summary, this project will provide health systems with a rigorous analysis of a defined set of tools to improve diabetes care for minority populations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus (based on fasting glucose, HbA1c, and problem list)
* At least 18 years old
* At least one face-to-face visit with Harvard Vanguard primary care clinician in the last 2 years

Exclusion Criteria:

* Any patient not categorized as either White or Black based on race identifier in the electronic medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Rate of LDL cholesterol control (< 100 mg/dL) | 12 months
Rate of blood pressure control (< 130/80 mmHg) | 12 months
Rate of HbA1c control (<7%) | 12 months

SECONDARY OUTCOMES:
Rate of HbA1c control (<8%) | 12 months
Rate of LDL cholesterol control (< 130 mg/dL) | 12 months
Rate of blood pressure control (< 140/90 mmHg) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Sequist, MD, MPH, Principal Investigator — Harvard Vanguard Medical Associates
Locations (1):
- Harvard Vanguard Medical Associates, Newton, Massachusetts, United States

REFERENCES:
- [Background] Sequist TD, Adams A, Zhang F, Ross-Degnan D, Ayanian JZ. Effect of quality improvement on racial disparities in diabetes care. Arch Intern Med. 2006 Mar 27;166(6):675-81. doi: 10.1001/archinte.166.6.675. PMID 16567608
- [Background] Sequist TD, Ayanian JZ, Marshall R, Fitzmaurice GM, Safran DG. Primary-care clinician perceptions of racial disparities in diabetes care. J Gen Intern Med. 2008 May;23(5):678-84. doi: 10.1007/s11606-008-0510-7. Epub 2008 Jan 24. PMID 18214625
- [Derived] Sequist TD, Fitzmaurice GM, Marshall R, Shaykevich S, Marston A, Safran DG, Ayanian JZ. Cultural competency training and performance reports to improve diabetes care for black patients: a cluster randomized, controlled trial. Ann Intern Med. 2010 Jan 5;152(1):40-6. doi: 10.7326/0003-4819-152-1-201001050-00009. PMID 20048271
- See also: HVMA website — http://www.harvardvanguard.org
- See also: Robert Wood Johnson Foundation national program office — http://www.solvingdisparities.org/